CLINICAL TRIAL: NCT04284566
Title: Effectiveness of a Multicomponent Treatment Based on Pain Neuroscience Education, Therapeutic Exercise, Cognitive Behavioural Therapy, and Mindfulness in Patients With Fibromialgia (FIBROWALK STUDY): A Randomized Controlled Trial
Brief Title: Effectiveness of Multicomponent Treatment for Fibromyalgia (FIBROWALK)
Acronym: FIBROWALK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Parc Sanitari Sant Joan de Déu (Other); Universitat Autonoma de Barcelona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FIBROWALK STUDY
Record Dates: First submitted 2020-02-23; First posted 2020-02-26 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Fibromyalgia
Keywords: multicomponent treatment; chronic pain; Fibromyalgia; pain neuroscience education; therapeutic exercise; cognitive behavioural therapy; mindfulness; randomized controlled trial
MeSH Terms: conditions — Fibromyalgia; Chronic Pain | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Single-blind, parallel-group, randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAU + multicomponent treatment FIBROWALK (Experimental): FIBROWALK is a multicomponent non-pharmacological program based on Pain Neuroscience Education (PNE), therapeutic exercise, Cognitive Behavioural Therapy (CBT) and Mindfulness Training
  Interventions: Behavioral: TAU + multicomponent treatment FIBROWALK
- Treatment as Usual (TAU) (Active Comparator): Treatment-as-Usual (TAU) consisted of prescribing drugs adapted to the symptomatic profile of each patient. The patients were instructed to continue their baseline medical treatment with no change throughout the 3-month period. In Spain, some counselling about aerobic exercise adjusted to patients' physical limitations is usually provided by first-line clinicians and specialists, but pharmacotherapy it's still the dominant treatment option. Patients were offered the opportunity to participate in the next wave of group intervention at the end of the study (3 months).
  Interventions: Behavioral: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: TAU + multicomponent treatment FIBROWALK — Group treatment protocol of 12 weekly 120 minute sessions. All sessions include the following ingredients (approx. in the same order):
  * Pain neuroscience education (30 min.)
  * Cognitive restructuring (30min.)
  * Mindfulness techniques (30 min.)
  * Physical exercise(30 min.)
  * Treatment as Usual (TAU) Standard pharmacological treatment usually provided to patients with fibromyalgia.
  Arms: TAU + multicomponent treatment FIBROWALK
Behavioral: Treatment as Usual (TAU) — Treatment-as-Usual (TAU) consisted of prescribing drugs adapted to the symptomatic profile of each patient. The patients were instructed to continue their baseline medical treatment with no change throughout the 3-month period. In Spain, some counselling about aerobic exercise adjusted to patients' physical limitations is usually provided by first-line clinicians and specialists, but pharmacotherapy it's still the dominant treatment option.
  Arms: Treatment as Usual (TAU)

SUMMARY:
The main objective of this study is to analyse the effectiveness of the FIBROWALK multicomponent treatment program as coadjuvant of treatment-as-usual (TAU) compared to TAU alone.

DETAILED DESCRIPTION:
This is a two-arm RCT focused on the potential efficacy of the multicomponent program FIBROWALK as coadjuvant of treatment-as-usual (TAU) vs. TAU alone. FIBROWALK combines multicomponent approach based on Pain Neuroscience Education (PNE), therapeutic exercise, Cognitive Behavioural Therapy (CBT) and Mindfulness training.

The main objective of this RCT was two-fold: (a) To analyse the effectiveness of a 12-week multicomponent treatment as an add-on to Treatment (FIBROWALK) as Usual (TAU) to improve functional impact (primary outcome), as well as pain, fatigue, kinesiophobia, physical function, anxiety, and depressive symptoms (secondary outcomes) compared to TAU; and (b) to explore the baseline differences between responders and non-responders in terms sociodemographic and clinical characteristics.

ELIGIBILITY:
Inclusion Criteria:

1. fulfil the 2010/2011 American College of Rheumatology (ACR) FM diagnostic criteria. The diagnosis was verified by a rheumatologist (MA) of the CSSSU
2. adults > 18 years old, and
3. provide written informed consent.

Exclusion Criteria:

1. To have a terminal illnesses or programmed interventions that might interrupt the study.
2. No stringent eligibility criteria were established due to the naturalistic nature of the RCT. Excluding patients with lower education or comorbidities might have turned away many patients from our RCT who would otherwise be eligible, that is we put emphasis on external validity. All recruited patients were considered capable of following the multicomponent therapy if they were allocated to it. Lack of adherence to drugs or home activities was not an exclusion criterion given the nature of our trial and we analysed data from all participants who underwent random allocation. Treatment allocation was performed by the clinical trials unit in accordance with computer-generated randomisation sequences.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-07-08 (Actual); Study Completion 2020-07-08 (Actual)

PRIMARY OUTCOMES:
Revised Fibromyalgia Impact Questionnaire (FIQR) | Through study completion, an average of 9 months
  The FIQR comprises three dimensions: physical dysfunction (scores from 0 to 30), overall impact (scores from 0 to 20), and intensity of the symptoms (scores from 0 to 50) is used to measure the impact generated by FM during the last week. It consists of 21 items, which are answered on a numerical rating scale of 11 points (from 0 to 10). Total scores can range from 0 to 100, with higher scores reflecting greater deterioration.

SECONDARY OUTCOMES:
Tampa Scale for Kinesiophobia (TSK-11) | Through study completion, an average of 9 months
  TSK-11 is used to assess fear of pain and movement. It consists of 11 items, which are answered on a Likert scale of 4 points. Total scores of each scale range from 11 to 44, where higher scores indicate a greater fear of pain and movement.
Visual Analog Scale (VAS) of the FIQR | Through study completion, an average of 9 months
  Visual Analog Scale (VAS) of the FIQR was used to measure fatigue and pain, with scores ranging from 0 to 10. Higher scores indicate greater perceived fatigue and pain, respectively.
Hospital Anxiety and Depression Scale (HADS) | Through study completion, an average of 9 months
  HADS is used to quantify the severity of anxiety and depression symptoms. It consists of two dimensions (anxiety and depression) of 7 items each responding on a Likert scale of 4 points. Total scores of each scale (HADS-A and HADSD) range from 0 to 21, where higher scores indicate greater severity of symptoms.
Physical Function of the 36-Item Short Form Survey (SF-36) | Through study completion, an average of 9 months
  Physical Function of the 36-Item Short Form Survey (SF-36) was used to measure physical function.This dimension comprises a total of 10 items, which are answered on a Likert scale of 3 points. Total scores on each scale are then transformed and can range from 0 to 100, with higher scores indicate better physical function.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Marsal, PhD, Study Chair — Vall d'Hebrón Hospital
Locations (1):
- Vall d'Hebrón Hospital, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Serrat M, Sanabria-Mazo JP, Almirall M, Muste M, Feliu-Soler A, Mendez-Ulrich JL, Sanz A, Luciano JV. Effectiveness of a Multicomponent Treatment Based on Pain Neuroscience Education, Therapeutic Exercise, Cognitive Behavioral Therapy, and Mindfulness in Patients With Fibromyalgia (FIBROWALK Study): A Randomized Controlled Trial. Phys Ther. 2021 Dec 1;101(12):pzab200. doi: 10.1093/ptj/pzab200. PMID 34499174